CLINICAL TRIAL: NCT06066658
Title: A Scoping Study to Evaluate the Potential of an Electronic Medical Device to Treat Anxiety in People Who Experience Breathlessness.
Brief Title: Anxiety Management in Breathlessness.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: LOROS Hospice Leicester (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0890
Record Dates: First submitted 2023-07-19; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-07

CONDITIONS: COPD; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Non randomised intervention and control both with standard care for breathlessness and anxiety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard care for Help with Breathlessness including medication, cognitive and behavioural strategies
- CES (Experimental): 8 weeks of 60 minutes a day 100microA a day with four week follow-up with standard care for help with breathlessness
  Interventions: Device: cranial electrotherapy stimulation (Alpha-Stim AID)

INTERVENTIONS:
Device: cranial electrotherapy stimulation (Alpha-Stim AID) — Alpha-Stim AID
  Arms: CES

SUMMARY:
The goal of this mixed methods study is to learn about cranial electrotherapy stimulation (CES) using Alpha-Stim AID in anxiety related to breathlessness in advanced lung diseases. The main question[s] it aims to answer are:

* Is CES using Alpha-Stim AID acceptable and tolerable as a potential treatment in the management of anxiety in patients who experience breathlessness due to advanced chronic respiratory disease?
* What are the key factors that will inform the design of a study to examine its potential clinical effectiveness? Participants will choose whether they want to trial the CES for eight weeks or be in a parallel control group. They will complete daily diaries, questionnaires about anxiety, breathlessness, sleep, quality of life and depression, and an end of study qualitative interview.

Researchers will compare those using the CES and those receiving standard care to see if there are any indications of difference in anxiety and other symptoms experienced.

DETAILED DESCRIPTION:
This is a two-site, mixed-methods, non-commercial interventional scoping study with a parallel non-randomised control group at LOROS Hospice (Leicester) and Northamptonshire Healthcare NHS Foundation Trust (NHFT) for patients with anxiety related to breathlessness secondary to advanced chronic respiratory disease.

Clinicians at both sites regularly complete the IPOS questionnaire as part of standard clinical practice. Patients who attend the HWB service will be screened for eligibility and approached by the research team for informed consent taking. Participants may choose to be in the intervention group or control group if places are available and the reasons for this choice will be noted in the CRF. This is in order to inform our feasibility objective for a future study.

Participants in the intervention group will receive an Alpha-Stim AID device with instruction on its use. The intervention is a single 60-minute session per day in their own home at a current of 100μA. This dose and/or duration of treatment may be modified at day 3 and/or day 5 in response to side effects as shown in the flowchart below (with a further review at day 7 if changes are made at day 5). Changes in the regime will be made after consultant with a medic (either CI or site PI).

The treatment period is 8 weeks, with a further 4 weeks of follow-up, totalling 12 weeks. The control group will be followed up for 12 weeks.

Demographic details and outcome measures will be recorded at baseline. A number of quantitative outcome measures will be collected in a daily log, at baseline, and weeks 2, 4, 8 and 12. Qualitative data via a semi-structured interview is sought from participants at the completion of the treatment and intervention period, or on withdrawal from either group unless due to significant clinical deterioration.

All participants will continue to receive standard care via their Hospice and their GP for the entirety of the study.

Inclusion criteria

* Aged 18 years or above. There is no upper age limit.
* Diagnosis of advanced chronic lung disease, including Chronic Obstructive Pulmonary Disease (COPD), Interstitial Lung Disease (ILD), or Pulmonary Fibrosis of any aetiology.
* Currently receiving care at LOROS or Northamptonshire Healthcare NHS Foundation Trust (NHFT)
* A score of 3 or 4 on IPOS Q2 for shortness of breath.
* A score of 2 or more on IPOS Q3 anxious or worried.
* Capable of giving oral and written informed consent to the study. Participants must be able to complete the validated outcome measures and daily log in English, however support from family can be utilised if English is not the participant's first language. Formal interpreters will be used for the consent and interviews if required.
* Agrees to return the Alpha-Stim AID device at the end of the study and not to purchase the device privately during the study.
* Estimated prognosis of >3 months at the time of recruitment.

Exclusion criteria

* Implantation with a pacemaker, cochlear implant, or an implantable cardioverter device (ICD).
* Neurological conditions, e.g. brain neoplasm, cerebrovascular events, epilepsy, neurodegenerative disorders, or prior brain surgery.
* Currently pregnant or planning a pregnancy.
* Involved with any other clinical trial at the time of consent.

Study procedures and assessments

Following informed consent, the IPOS questionnaire will be completed if required as further eligibility screening. Eligible participants will then complete baseline measurements:

* Demographics and clinical characteristics, including age, gender, ethnicity, primary diagnosis of chronic respiratory disease, and current medication (both acute and repeat prescriptions).
* GAD-7 (Spitzer et al, 2006).
* CRQ-SR (Williams et al, 2001).
* D-12 (Yorke et al, 2010).
* Sleep Condition Indicator (Espie et al. 2014).
* PHQ-9 (Kroenke, Spitzer, and Williams, 2006).
* EQ-5D-5L (EuroQol group, 2017).
* Participants will also be asked to complete the 0-10 NRS scales in the daily log at the end of day 1.

The baseline assessment/screening will be undertaken by a researcher or research nurse and inputted into the trial database.

Participants in the treatment group will be given an Alpha-Stim AID device and trained in its use. They will be asked to note each day in their daily log how long they used the device for and the nature and severity of any side effects they are experiencing.

All participants will be asked to complete the NRS for anxiety and breathlessness for the day in their daily log. All participants will be encouraged to add free text comments to their daily log to reflect their experience of breathlessness, anxiety and any changes in this.

Questionnaire Outcome measures will be repeated at 2,4, 8 and 12 weeks

Participants will receive a phone call or text message 2 days in advance of when the outcome measure is due to be collected to arrange a study face to face visit or to determine their preferred method for questionnaire completion (either with the assistance of a researcher/research nurse or independently to then return in a stamped addressed envelope to LOROS). If a response is not received within 2 days, a second attempt at contact will be made, and a third 2 days thereafter. Participants will not be accepted as lost to follow-up until three attempts at contact have been made. Data collected from those who are lost to follow up will be retained and this will be outlined in the participant information sheet.

All participants will be seen face to face at their hospice (either LOROS or Northamptonshire Healthcare NHS Foundation Trust) or within their homes), whichever is preferred by the participant, at baseline, week 2 and week 12. Researchers will follow the lone worker policy of their own employing organisations. If participants incur any travel expenses as a result of their participation these may be reimbursed on production of a receipt for public transport or as a claim for mileage which would be reimbursed at LOROS. Reasonable travel expenses will be paid in full.

At week 4 all participants may choose a face to face or virtual study contact. At week 8 participants in the intervention group will be seen face to face (end of treatment), those in the control group can choose face to face or virtual study contact.

If participants are unable to be seen face to face, for example if they contract COVID, then these meetings can be carried out virtually via video or telephone call.

Contact will be made with participants in the intervention group by phone, text or email (as per their preference) on day 3 and day 5 to assess adverse effects and support the participant in use of the device and make changes in the duration or dose as required. If a change is made a further contact will be made 2 days later. Notes will be made in the CRF about adverse effects, change in intervention and support provided.

The semi-structured interview at the end of the study or at withdrawal may be face to face or via phone or video call as preferred by the patient. Face-to-face meeting may be at the Hospice or in the participants' own home as preferred. Interviews may take place up to 2 weeks after the completion of the study period as per the participant's availability.

The GP (by letter) and the Hospice clinical team (by recording in the patients' notes) will be informed of patients' involvement in the study. Researchers will liaise with the patient's Hospice clinical team to ensure that all ongoing contact is sensitive, seeking to know if patients have died or significant deterioration has occurred that may impact on their continuation in the study.

Qualitative assessments The daily log will comprise of two pages to complete each day for the intervention group, and one page each day for the control group. Participants will be asked to complete the three NRS 0-10 scales for both anxiety and breathlessness each day. For the treatment group, there will also be a space to record the usage of the Alpha-Stim AID device and any side effects they may be experiencing. Each daily entry will also include a space to record the use of any PRN medications for anxiety and breathlessness, as well as an area for free text comments. Participants will be encouraged to complete this free text area with information about why they have given the 0-10 NRS scores for that day, their thoughts on the treatment, or any other comments they want the researchers to know.

At the end of the 8 week intervention period, participants will be asked to reflect on their use of the Alpha-Stim AID over 8 weeks in the daily log and/or verbally to the researcher. Comments will be noted in the CRF.

The daily logs will be checked at week 2 to ensure that the participants are able to complete them correctly, and collected at each face to face contact point or in full at the end of the study period. Free text comments will be collected as qualitative data.

Semi-structured interviews will take place at the end of the study period or if participants withdraw (unless due to significant clinical deterioration). The interviews will explore participants' lived experience of breathlessness anxiety over the study period. For the treatment group, we also aim to explore their thoughts and opinions on the Alpha-Stim AID device and participation in the study. It is important for the researchers to also understand qualitatively if participants describe feeling any different than at baseline, in order to correlate this with our patient-reported outcome measures. We will explore barriers and facilitators to using CES in order to improve our study for a potential larger scale trial in the future. This will allow us to meet our primary objective of measuring the acceptability and feasibility of CES in our target population.

The interviews will be conducted either via phone, video-call, or face-to-face, depending on COVID-19 measures and patient preference. Interviews will be carried out by experienced researchers associated with NHFT and LOROS Hospice and will be recorded on a password protected recorder. Audio files will be stored on an encrypted computer and deleted once they have been transcribed Interviews will be one-to-one unless the participant requests the support of their family or requires an interpreter. A local interpreting service which has been utilised by UoL and LOROS hospice previously will be used where needed. The interpreters will be briefed about the study and their involvement prior to each interview. They will also be debriefed post-interview to capture any additional information. The interpreters/interpreting service will sign standard UoL/LOROS contracts and confidentiality agreements as necessary. We will work with the interpreting service to provide quality assurance.

If a response is not received within 3 days, a second attempt at contact will be made, and a third 3 days thereafter. The qualitative component of the study is not an optional aspect of the design.

Sample size This is a scoping study to understand a number of feasibility factors pertinent to study design that are hitherto unknown. The sample size chosen is also related to the resources available. We will recruit participants over 9 months.

We estimate based on historical data that in 9 months at least 60 patients would be seen across the two recruitment sites that meet the eligibility criteria. From previous studies in palliative care we estimate that 50% of people would agree to participate and that 60% would complete the 12 week study period (40% attrition). However these recruitment, completion/attrition parameters in the specific context of anxiety and breathlessness and the trial of the alpha-stim device are unknown and ascertaining them is a key aspect of the study.

We have therefore adopted an unusual design of an unknown recruitment sample size which will aim to achieve 10 participants completing in each arm of the study. We estimate that this will require approaching 60 people, and consenting 30 participants. Eligibility, acceptability and attrition will all affect the sample size that is finally recruited.

We will aim to recruit participants to the intervention group over a staggered period of nine months in order to closely observe and support each participant. A sample of 10 completing treatment and trial measures together with any who withdraw from the study is likely to give sufficient qualitative and quantitative data to understand the primary objective for the study (acceptability and safety).

A quantitative data set for 20-30 participants (both control and treatment) will give a good basis for understanding how outcome measures change over time and participant feedback on the measures and will inform future questions and study design. It may give some indications of potential for effectiveness but the sample size is not designed to establish this.

The sample size will report recruitment rates with 95% precision for confidence interval of around 36%. The ease and rate of recruitment and attrition/completion rates in this scoping study will help guide the sample size and recruitment rate and number of sites required for recruitment for a future larger study if appropriate.

Statistical methods Descriptive analysis of quantitative measures will be conducted.

Primary outcome analysis Daily log data will be used to evaluate and describe level of compliance with the standard regime of 60-minutes 100uA or with the personalised regimes B and C.

The key analysis is % of participants fully complying with their given regime. Other analysis will involve the mode and range of frequency (how many days out of 7) and duration (how many minutes) of use.

Daily log data will be used to quantify type, number, severity and duration of adverse effects.

Secondary outcome analysis Percentages and descriptive statistics will be used to summarise the secondary outcomes.

Tertiary and quaternary outcome analysis The change over time for outcome measure (NRS-anxiety, NRS-breathlessness, GAD-7, CRQ-all domains, D-12, PHQ-9, SCI, IPOS and EQ-5D-5L) will be described and plotted for the treatment and control groups and compared in graphical plots of participant scores to assess the potential that treatment has had an impact.

Analysis of qualitative data Analysis of the qualitative data from interviews and daily logs will begin with manual transcription of the interview audio files and the collection of each participant's daily log entries into a Word document.

The transcriptions and daily log entries will each be coded. Codes will then be grouped into themes in a process of inductive thematic analysis, where themes emerge from the data rather than being constructed from a pre-defined hypothesis. Researchers will practice reflexivity throughout the entire analysis process. The initial 15% of interviews will be coded by two researchers simultaneously but independently of each other. Discrepancies will then be reviewed by the CI and adjustments made accordingly. The remainder of the interviews will be coded by a single researcher. Qualitative analysis software will support the data analysis.

Data from notes in CRFs will be integrated with our sources of information to address the feasibility questions

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above. There is no upper age limit.
* Diagnosis of advanced chronic lung disease, including Chronic Obstructive Pulmonary Disease (COPD), Interstitial Lung Disease (ILD), or Pulmonary Fibrosis of any aetiology.
* Currently receiving care at LOROS or Cynthia Spencer Hospice.
* A score of 3 or 4 on IPOS Q2 for shortness of breath.
* A score of 2 or more on IPOS Q3 anxious or worried.
* Capable of giving oral and written informed consent to the study.
* Agrees to return the Alpha-Stim AID device at the end of the study and not to purchase the device privately during the study.
* Estimated prognosis of >3 months at the time of recruitment.

Exclusion Criteria:

* Implantation with a pacemaker, cochlear implant, or an implantable cardioverter device (ICD).
* Neurological conditions, e.g. brain neoplasm, cerebrovascular events, epilepsy, neurodegenerative disorders, or prior brain surgery.
* Currently pregnant or planning a pregnancy.
* Involved with any other clinical trial at the time of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability and tolerability | 2,4,8 and 12 weeks
  qualitative text entries in daily log and analysis of end of study interviews will be triangulated with adverse effects (number of participants experiencing AE thought to be causally related to the CES, severity, and duration) and in comparison to those in control arm. We do not anticipate SAE to be a feature of the study.

SECONDARY OUTCOMES:
Anxiety | baseline, 2, 4, 8 and 12 weeks
  using GAD 7 (General Anxiety Disorder) This is a validated, widely used 7 item questionnaire with frequency of experience over the past two weeks categories (not at all, several days, over half the days and nearly every day

CONTACTS AND LOCATIONS:
Overall Officials: christina faull, MBBS, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - LOROS Hospice, Leicester, Leicestershire
  - Northamptonshire Healthcare NHS Trust, Northampton

IPD SHARING:
Plan to Share IPD: No